CLINICAL TRIAL: NCT00560976
Title: Serum Neutrophil Gelatinase Associated Lipocalin (NGAL) Levels in Hemodialysis (HD) Patients; Relation to Iron Status, Hemodialysis, and Intravenous (IV) Iron Administration
Brief Title: Serum NGAL Levels in Hemodialysis (HD) Patients; Relation to Iron Status, HD and Intravenous (IV) Iron Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, David Tovbin, Dr David Tovbin, Department of Nephrology, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor419105ctil
Record Dates: First submitted 2007-11-18; First posted 2007-11-20 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: neutrophil gelatinase associated lipocalin; hemodialysis; iron; inflammation; Oxidative Stress
MeSH Terms: conditions — Inflammation | interventions — Ferric Oxide, Saccharated; ferric gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron Saccharate (Venofer) (Experimental): IV Iron Saccharate (Venofer)100 mg
  Interventions: Drug: Iron Saccharate (Venofer)

INTERVENTIONS:
Drug: Iron Saccharate (Venofer) — Hemodialysis with IV iron administration of 100 mg Iron Saccharate (Venofer) in 150 ml 0.9 % saline to the arterial dialysis line during first hour of mid-week dialysis session. An alternative IV iron brand in some centers participating in the study could bebe 62.5 mg ferric gluconate (Ferrlecit).
  Other Names: Ferric gluconate (Ferrlecit)

SUMMARY:
The purpose of this study is to assess changes in serum levels of the siderophore binding protein NGAL by hemodialysis without and with intravenous iron administration

DETAILED DESCRIPTION:
Serum and urine levels of the siderophore binding protein neutrophil gelatinase associated lipocalin (NGAL) are increased in a number of renal diseases, but has not been evaluated yet in dialysis patients. Since NGAL is suggested to be related to inflammatory processes and iron homeostasis, which are a major problem in dialysis patients, this study aims to assess the relation of serum NGAL levels in hemodialysis (HD) patients to iron status, inflammation, hemodialysis and intravenous(IV) iron administration. Our hypothesis is that serum NGAL levels in HD patients are related to iron status and inflammation and may change following hemodialysis and/or acute or chronic IV iron administration.

The Specific aims are:

1. To assess the relations between basal serum NGAL levels to iron, dialysis, and inflammation related parameters.
2. To assess the effect of HD on serum NGAL levels and their relation with with iron, dialysis and inflammation related parameters.
3. To assess the effects of weekly 100 mg IV iron in the first hour of HD on serum NGAL levels, and the relation of pre IV iron serum NGAL levels with iron, oxidative stress and inflammation related parameters. These assessments will be performed in the first weekly HD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients

Exclusion Criteria:

* Acute disease (infection, thrombosis, ischemia, bleeding)
* Hepatitis B, Hepatitis C or HIV
* Intravenous iron administration or packed red cell transfusion in the last 4 weeks prior to the study

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
CRP (C-Reactive Protein) and AOPP (Advanced Oxidative Protein Products) Levels | To assess the effects of 100 mg IV iron in the first hour of the first weekly HD on the relation of pre IV iron serum NGAL levels with oxidative stress and inflammation related parameters.

CONTACTS AND LOCATIONS:
Overall Officials: David Tovbin, MD, Principal Investigator — Soroka University Medical Center
Locations (3):
- Israel (3):
  - Department of Nephrology, Soroka University Medical center, Beersheba
  - Bnai-zion Medical Center,Nephrology,, Haifa
  - Department of Nephrology, Wolfson Medical Center, Holon